CLINICAL TRIAL: NCT02184247
Title: A Study to Compare the Bioavailability of Two Sustained-release Theophylline Products
Brief Title: Bioavailability of Two Sustained-release Theophylline Products in Healthy Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1071.10
Record Dates: First submitted 2014-07-08; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Theophylline

ARMS (2):
- anhydrous theophylline, 350 mg (Experimental)
  Interventions: Drug: anhydrous theophylline, 350 mg
- anhydrous theophylline, 300 mg (Active Comparator)
  Interventions: Drug: anhydrous theophylline, 300 mg

INTERVENTIONS:
Drug: anhydrous theophylline, 350 mg
  Other Names: Bronchoretard®
  Arms: anhydrous theophylline, 350 mg
Drug: anhydrous theophylline, 300 mg
  Other Names: Theo-Dur®
  Arms: anhydrous theophylline, 300 mg

SUMMARY:
Study to compare the bioavailability of 350 mg Bronchoretard® - a sustained-release theophylline (anhydrous) product with respect to the reference product, Theo Dur® 300 mg theophylline anhydrous (sustained-release product) by comparing the rate and extent of absorption of theophylline based on both single and multiple-dose profiles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-smoking male subjects between 18 and 45 years of age
* Body weight within 10% of the ideal weight according to the Body Mass Index (BMI)
* Normal health based on medical history and findings within the range of clinical acceptability, in respect of the physical examination (including electrocardiogram and vital signs) and special investigations
* Ability to comprehend and willingness to sign both statements of informed consent (for screening and study-specific procedures)

Exclusion Criteria:

* History of serious systemic or organ disease
* A major illness during the 3 months before commencement of the study-related procedures
* Significant physical or organ abnormality
* History of hypersensitivity to theophylline or other xanthine derivatives
* Use of any medication within 2 weeks before the first administration of study medication
* Participation in another study with an experimental drug within 8 weeks before the first administration of study medication
* Treatment within the previous 3 months with any drug with a well-defined potential for adversely affecting a major organ or system (for example chloramphenicol, which may cause bone marrow suppression)
* Donation of blood during the 8 weeks before the first administration of study medication
* History of, or current compulsive alcohol abuse (> 10 drinks per week), of regular exposure to other substance of abuse
* Positive testing for HIV and hepatitis B antigens within the previous 3 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 1998-04; Primary Completion 1998-05 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | up to 36 hours after first drug administration
Area under the plasma concentration versus time data pairs, with extrapolation to infinity (AUDC) | up to 36 hours after first drug administration
Area under the plasma concentration versus time data pairs at steady state (AUDss) | up to 12 hours after last administration of study drug
Percent peak-to-trough fluctuation (%PTF) | up to 12 hours after last administration of study drug

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | up to 36 hours after first drug administration
Apparent terminal half-life (t1/2.z) | up to 36 hours after first drug administration
Area under the plasma concentration versus time data pairs [AUD(0-tlast)], also indicated by AUD, where tlast is the time of the last quantifiable concentration | up to 36 hours after first drug administration
Ratio of Cmax and AUDC (Cmax/AUDC) | up to 36 hours after first drug administration
Total mean time in the system (MTvsys) | up to 36 hours after first drug administration
Maximum concentration at steady state (Cmax,ss) | up to 12 hours after last administration of study drug
Minimum concentration at steady state (Cmin,ss) | up to 12 hours after last administration of study drug
Plateau time (T75%Cmax) | up to 12 hours after last administration of study drug